CLINICAL TRIAL: NCT04326803
Title: Hepatitis B Virus (HBV) Infection in Haitian Immigrants in Chile: Determination of HBV Genotypes, Viral Escape Mutants and Host Factors Influencing Response to Vaccination
Brief Title: Hepatitis B en Haitian Immigrants in Chile: Molecular Characterization and Determination of Vaccine Response
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 180814005; 1191389 (Other Grant/Funding Number: FONDECYT (Chile))
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Hepatitis B
Keywords: hepatitis B; migration; HIV
MeSH Terms: conditions — Hepatitis B | interventions — COMVAX

STUDY DESIGN:
Intervention Model Description: A single group of subject will be offered to enroll in a study to assess the serological response to an accelerated schedule (0, 1 and 6 months) of recombinant hepatitis B vaccine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vaccine group (Experimental): Administration of 3 doses hepatitis B vaccine (recombinant hepatitis B vaccine, injectable suspension for intramuscular use) at month 0, 1 and 2.
  Interventions: Biological: Hepatitis B recombinant vaccine

INTERVENTIONS:
Biological: Hepatitis B recombinant vaccine — Administration of 20 mcg of hepatitis B recombinant vaccine im at month 0, 1 and 2
  Other Names: Engerix-B vaccine

SUMMARY:
International migration to Chile has sharply increased since 2010. Particularly, Haitian migration now totals approximately 200.000 people. Preliminary results show a high prevalence of hepatitis B infection in this population. Approximately 35% of adult Haitian migrants in Chile have been exposed to hepatitis B infection. In this study the investigators aim to study the clinical and molecular characteristics of this infection and also to assess the serological response to an accelerated schedule of hepatitis B vaccination (0, 1 and 2 months).

DETAILED DESCRIPTION:
Migration from Haiti to Chile has increased exponentially in the last years. More than 200.000 people from this island are currently living in Chile. Preliminary results of the investigators group show that HIV infection and hepatitis B virus (HBV) infection are 2.9% and 2.4% (14 and 16 times higher than the reported prevalence in Chile), respectively, and overall HBV infection (anti-HBc antibody) is 34%. The molecular characterization of the HBV variants infecting people from Haiti has not been carried out. The current evidence suggests that HBV traveled from Africa together with the slave trade 200 to 300 years ago, with genotypes infecting Haitians resembling that of their origins, but with some striking differences, such as the presence of a recently described subtype (A5), which is now uncommon in Africa. HBV genotypes and subgenotypes may influence the emergence of specific mutations in the surface antigen region of the virus which in turn could lead to escape mutants which can infect properly vaccinated people. There is no information regarding the genotypes and escape mutants in Haitian immigrants to Chile. The most effective way to control and prevent is vaccination, but the response to vaccination varies widely in different ethnic groups, with genetic factors being relevant. Mutations in the interferon lambda 3 gene (IFNL3), previously known as interleukin 28B (IL28B) are clearly associated with lower response to interferon treatment and spontaneous clearance in hepatitis C, and clinical evolution of various viral infections. Less favorable IFNL3 mutations are especially prevalent in African descendants. The hypothesis of the project is that Haitian immigrants in Chile have a high prevalence of HBV infection with viral genotypes/mutations different from the native Chilean genotypes, which may result in a particular clinical presentation. The investigators also conjecture that the response to HBV vaccination may also differ in Haitian immigrants due to genetic variations in the IFNL3 gene. The HBV infection prevalence in this population will be estimated and the researchers will try to explain if mutations in IFNL3 increase the rate of spontaneous clearance of the infection (comparing carriers to patients who cleared the infection). They will also determine the presence of HBV DNA in all enrolled subjects to study the occurrence of occult hepatitis B (OBI), which is the presence of DNA in the absence of HBsAg. HBV DNA will be amplified and sequenced in the pre-S1, pre-S2 and S region (surface antigens) to study the presence of escape mutants. Finally, the investigators will conduct a study of vaccination of Haitian immigrants to assess the effectiveness of the vaccine in this population and determine which factors may influence vaccine response, including mutations in the IFNL3 gene. The information regarding the prevalence, epidemiology, presence of escape mutants, genetic factors influencing HBV infection and the response to the vaccine in Haitian immigrants, are critical for a better understanding of this infection and for the development of public health policies based on scientific evidence and not in political or other reasons that usually perpetuate stigma and inequalities in health care for marginalized groups.

ELIGIBILITY:
Inclusion Criteria:

* Adults (> 18 yo) born in Haiti.
* Living in Chile (and planning to stay in Santiago for the next 4 months).

Exclusion Criteria:

* Not signing the informed consent.
* Pregnancy.
* HIV or HCV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Response rate | 4-8 weeks after the third dose of the vaccine
  Developing antibodies against HBsAg (anti-HBs) > 10 mIU/mL

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Soza, MD, Principal Investigator — Pontificia Universidad Catolica de Chile

IPD SHARING:
Plan to Share IPD: No
Available on request

REFERENCES:
- [Background] Zampino R, Boemio A, Sagnelli C, Alessio L, Adinolfi LE, Sagnelli E, Coppola N. Hepatitis B virus burden in developing countries. World J Gastroenterol. 2015 Nov 14;21(42):11941-53. doi: 10.3748/wjg.v21.i42.11941. PMID 26576083
- [Background] Locarnini S, Hatzakis A, Chen DS, Lok A. Strategies to control hepatitis B: Public policy, epidemiology, vaccine and drugs. J Hepatol. 2015 Apr;62(1 Suppl):S76-86. doi: 10.1016/j.jhep.2015.01.018. PMID 25920093
- See also: Site in Spanish with information about viral hepatitis and liver diseases. — http://hepatitis.cl